CLINICAL TRIAL: NCT02824926
Title: Non-inferiority Phase II Trial Comparing BL123 (Biolab Sanus Farmacêutica Ltda.) Versus Ketoconazole (Nizoral® Janssen-Cilag) in Patients With Tinea Pedis
Brief Title: Clinical Trial Comparing BL123 Versus Ketoconazole in Patients With Tinea Pedis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilberto De Nucci (Other Government)
Collaborators: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor-Investigator, Gilberto De Nucci, PhD, Galeno Desenvolvimento de Pesquisas Clínicas
Organization: Galeno Desenvolvimento de Pesquisas Clínicas (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDN 083/13
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis | interventions — 1-(2-(2,4-dichlorophenyl)-2-(4-(trifluoromethyl)benzyloxy)ethyl)-1H-imidazole; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapaconazole (Experimental): (cream; 2%; topical)
  Interventions: Drug: Dapaconazole
- Ketoconazole (Active Comparator): (cream; 2%; topical)
  Interventions: Drug: Ketoconazole

INTERVENTIONS:
Drug: Dapaconazole
  Arms: Dapaconazole
Drug: Ketoconazole
  Arms: Ketoconazole

SUMMARY:
This is a non-inferiority, Phase II, open-label, randomized, parallel trial to evaluate efficacy and safety of the new intervention (Dapaconazole cream 2%) versus the active control (Ketoconazole cream 2%) in patients with Tinea Pedis. Study schedule comprises enrollment, treatment and follow-up visits. Treatment period is 14 days.

DETAILED DESCRIPTION:
The study sample consists of male and female subjects aged between 18 and 60 years-old, either with single or multiple Tinea Pedis lesion(s). Sixty (60) patients will be enrolled, but each foot with lesion(s) will be considered as one (1) sample. Therefore, if a patient has bilateral lesions, one foot will be allocated to investigational product (Dapaconazole) and the other foot will be allocated to active control (Ketoconazole). Randomization will determine which foot (right or left) will be treated with Dapaconazole or Ketoconazole.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 18 and 60 years-old;
* Presence of skin lesion(s) characteristic of Tinea Pedis, with diagnosis confirmed by direct mycological exam;
* Absence of previous antifungic treatment for the current lesion(s) under study;
* Absence of other significant diseases which, at physician's discretion, could have an impact on subject's participation in the trial, according to protocol requirements and study evaluations: medical history, blood pressure and heart rate, physical examination and screening laboratory tests;
* Ability to understand the nature and objectives of the trial, including its risks and adverse events; willingness to cooperate with the researcher and proceed according to all study requirements, which shall be confirmed by Informed Consent Form signature.

Exclusion Criteria:

* Known hypersensitivity to ketoconazole or chemically related compounds; history of serious adverse reactions;
* Current evidence of clinically significant diseases which, at physician's discretion, prevent subject's participation in the trial and/or expose the subject to risks other than what is normally expected;
* Use of medications that, at principal investigator's discretion, might expose the subject to risks other than what is normally expected;
* Screening laboratory tests results showing clinically relevant deviations that, due to potential risks, prevent participation in the trial, at the researcher's discretion;
* Drugs addiction, including alcohol;
* Use of any previous treatment to the lesion(s) under study that, according to principal investigator's discretion, might interfere with the study objectives;
* Treatment, within 3 months before this trial, with any drugs known to have a well-established toxic potential to major organs;
* Participation in any other experimental research or administration of any experimental drug within 6 months before this trial;
* Positive pregnancy test, labor or miscarriage within 12 weeks before study treatment;
* Any conditions, according to investigator's discretion, that prevent subjects to participate in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Clinical cure of the lesion(s) | 14 days
  Assessment of presence or absence of lesion(s) by clinical examination
Mycological cure of the lesion(s) | 14 days
  Laboratory test for presence or absence of Tinea Pedis

SECONDARY OUTCOMES:
Time (days) to clinical diagnosis of lesion(s) cure | 14 days
Time (days) to absence of itching at lesion(s) site | 14 days

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 45 days
  Number of adverse events
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 45 days
  Changes of laboratory parameters that are out of normal values/ranges and/or considered as clinically significant by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, PhD, Principal Investigator — Galeno Desenvolvimento de Pesquisas Ltda.

IPD SHARING:
Plan to Share IPD: Yes
No IPD available.